CLINICAL TRIAL: NCT01279174
Title: Whole Body Vibration Compared to Conventional Physiotherapy in Patients With Coxarthrosis: a Randomized, Controlled Study
Brief Title: Galileo-Hip Whole Body Vibration /Conventional Physiotherapy /Coxarthrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Kourosh Zarghooni, Dr.med., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ortho-Koeln-1-2011; Version V1.55 (Other Grant/Funding Number: P228 A57 Eysel EP2 hüfte Ko I 21 k 2010 12)
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Coxarthrosis
Keywords: Hip, arthrosis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional physiotherapy (Other): Patients in this study group will attend physiotherapeutic exercise sessions of one hour three times a week for six weeks. The sessions consist of aerobic and muscle strengthening as well as coordination exercises. Patients will practice activities of daily living. The goals of these exercises are to improve joint stability, optimize knee and ankle proprioception, and advance neuromuscular innervation of the lower extremity and thereby suppress pathologic motion patterns. This should lead to optimized mobility, increased stability, and thus more endogenous analgesia of the affected joint
  Interventions: Other: Conventional physiotherapy
- Whole-body-vibration exercises (Experimental): Patients in this study group will attend whole body vibration exercise sessions of one hour three times a week for six weeks, using the Galileo® Fitness device. Initial training sessions will focus on patient acclimatization, and afterwards improved on muscular capacity and body coordination. During exercise sessions, patients will do 6 training cycles of 3 minutes each. The goals of this treatment are improved proprioception of the ankle and knee joints, as well as optimization of neuronal reactivation of the muscles and thereby improved joint stability. This should also increase endogenous analgesia
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: Conventional physiotherapy — Patients in this study group will attend physiotherapeutic exercise sessions of one hour three times a week for six weeks. The sessions consist of aerobic and muscle strengthening as well as coordination exercises. Patients will practice activities of daily living. The goals of these exercises are to improve joint stability, optimize knee and ankle proprioception, and advance neuromuscular innervation of the lower extremity and thereby suppress pathologic motion patterns. This should lead to optimized mobility, increased stability, and thus more endogenous analgesia of the affected joint

SUMMARY:
Osteoarthritis (OA) is the most common degenerative arthropathy. Load-bearing joints such as knee and hip are more often affected than spine or hands. The prevalence of gonarthrosis is generally higher than that of coxarthrosis.

Because no cure for OA exists, the main emphasis of therapy is analgesic treatment through either mobility or medication. Non-pharmacologic treatment is the first step, followed by the addition of analgesic medication, and ultimately by surgery.

The goal of non-pharmacologic and non-invasive therapy is to improve neuromuscular function, which in turn both prevents formation of and delays progression of OA. A modification of conventional physiotherapy, whole body vibration has been successfully employed for several years. Since its introduction, this therapy is in wide use at our facility not only for gonarthrosis, but also coxarthrosis and other diseases leading to muscular imbalance.

DETAILED DESCRIPTION:
This study is a randomized, therapy-controlled trial in a primary care setting at a university hospital. Patients presenting to our outpatient clinic with initial symptoms of coxarthrosis will be assessed against inclusion and exclusion criteria. After patient consent, 6 weeks of treatment will ensue. During the six weeks of treatment, patients will receive one of two treatments, conventional physiotherapy or whole-body-vibration exercises of one hour three times a week. Follow-up examinations will be performed immediately after treatment and after another 6 and 20 weeks, for a total study duration of 6 months. 20 patients will be included in each therapy group.

ELIGIBILITY:
Inclusion Criteria:

* Age 30 - 80 years
* Body weight less than or equal to 160 kg
* Body-Mass-Index less than 40 kg/m²
* Outpatient
* Legal competence
* Signed informed consent
* Uni- or bilateral Coxarthrosis according to ACR criteria
* WOMAC-pain index (visual analogue scale) of 30-70 mm
* Coxarthrosis stage II-III according to Kellgren and Lawrence

Exclusion Criteria:

* Participation in parallel interventional studies
* Bilateral Coxarthrosis with WOMAC Pain index more than 70 mm
* Previous surgery during the past 6 months at the Index Joint
* Injury of the study joint during the last 6 months
* Secondary rheumatoid or septic arthrosis or systemic diseases affecting the study joint
* Activated coxarthrosis with intraarticular effusion
* Body weight > 160 kg or body mass index > 40 kg/m²
* Analgesic therapy with steroidal drugs
* Physiotherapy of the lower extremities during the past 6 weeks
* Existing endoprosthetics in the lower extremities

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Changes in Womac | 26 weeks
  The primary outcome measure is the patients' evaluation of improvement on the visual analogue scale of the WOMAC indices for pain and activities of daily life, comparing baseline and post-treatment. The secondary outcome measures summarized in the appendices will also be assessed at baseline and after 6, 12, and 26 weeks

SECONDARY OUTCOMES:
SF-12 | 26 weeks
  The SF-12 score uses subjective patient responses to measure success of therapy and thereby evaluate quality of life. SF-12 is the abbreviated version of the SF-36 Health Survey and contains 12 items representing 8 dimensions of physical and mental fitness. In our study, the validated German translation will be used
Leonardo Mechanography | 26 weeks
  Functional motion analysis, the Modified Clinical Test of Sensory Interaction in Balance, the Tandem Walk Test, and the Rhythmic Weight Shift Test will be performed using the Leonardo Mechanography Gangway (Novotec Inc., Pforzheim, Germany) and the Balance Master Analysis System (Neurocom Inc., Clackamas, USA). These will provide reliable data on essential parts of ambulation, e.g. stride length, speed of movement, shifting of balance point, force, power, and workload

CONTACTS AND LOCATIONS:
Overall Officials: Peter Knöll, Principal Investigator — University Hospital of Cologne
Locations (1):
- University Hospital, Cologne, Germany